CLINICAL TRIAL: NCT03156218
Title: The Effect of Inspiratory Oxygen Fraction on the Ratio of Partial Arterial Oxygen Pressure and Inspiratory Oxygen Fraction (PaO2/FiO2 Ratio) in Mechanically Ventilated Patients With and Without Mild to Moderate ARDS
Brief Title: The Effect of FiO2 on PaO2/FiO2 Ratio
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Amsterdam UMC, location VUmc (Other)
Responsible Party: Principal Investigator, Angelique Spoelstra-de Man, Principal Investigator, Amsterdam UMC, location VUmc
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: NL61945.029.17
Record Dates: First submitted 2017-05-15; First posted 2017-05-17 (Actual); Last update posted 2019-04-26 (Actual); Status verified 2019-04

CONDITIONS: PaO2/FiO2 Ratio
Keywords: PaO2/FiO2 ratio, hyperoxia, mechanical ventilation, ARDS
MeSH Terms: conditions — Hyperoxia

STUDY DESIGN:
Intervention Model Description: In both groups FiO2 will be modulated: FiO2 will be reduced to 21% or until peripheral oxygen saturation of 92%, whatever occurs first. Subsequently FiO2 will be increased up to 100%.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Without ARDS (Experimental): Patients admitted to the ICU after cardiac surgery with a PaO2/FiO2 ratio > 300.
  Modulation of FiO2: FiO2 will be reduced to 21% or until peripheral oxygen saturation of 92%, whatever occurs first. Subsequently FiO2 will be increased up to 100%.
  Interventions: Drug: Modulation of FiO2
- With mild to moderate ARDS (Experimental): Patients admitted to the ICU after cardiac surgery with a PaO2/FiO2 ratio > 100 and < 300.
  Modulation of FiO2: FiO2 will be reduced to 21% or until peripheral oxygen saturation of 92%, whatever occurs first. Subsequently FiO2 will be increased up to 100%.
  Interventions: Drug: Modulation of FiO2

INTERVENTIONS:
Drug: Modulation of FiO2 — Modulation of FiO2: FiO2 will be reduced to 21% or until peripheral oxygen saturation of 92%, whatever occurs first. Subsequently FiO2 will be increased up to 100%.

SUMMARY:
The PaO2/FiO2 ratio is frequently used to determine the severity of lung injury in mechanically ventilated patients. However, several mathematical models have shown that PaO2/FiO2 ratio depends on FiO2. The relationship is complex and depends on numerous physiological variables, including shunt fraction, and arterio-venous oxygen difference. The nonlinear relation between PaO2/FiO2 and FiO2 underlines the limitations describing the intensity of hypoxemia using PaO2/FiO2 and is thus of major importance for the clinician. Surprisingly, this relationship has only been assessed mathematically. Obviously, the accuracy of the mathematical relationship depends on the input variables used.

The current study is designed to assess the PaO2/FiO2 vs FiO2 relation in mechanically ventilated patients without ARDS (n =10) and with mild or moderate ARDS (n =10). In order to explain the dependency of the PaO2/FiO2 on FiO2, shunt fraction and alveolar - arterial oxygen difference ((A-a)DO2) will be determined in these patients.

DETAILED DESCRIPTION:
Rationale:

The PaO2/FiO2 ratio is frequently used to determine the severity of lung injury in mechanically ventilated patients. However, several mathematical models have shown that PaO2/FiO2 ratio depends on FiO2. The relationship is complex and depends on numerous physiological variables, including shunt fraction, and arterio-venous oxygen difference. The nonlinear relation between PaO2/FiO2 and FiO2 underlines the limitations describing the intensity of hypoxemia using PaO2/FiO2 and is thus of major importance for the clinician. Surprisingly, this relationship has only been assessed mathematically. Obviously, the accuracy of the mathematical relationship depends on the input variables used.

The current study is designed to assess the PaO2/FiO2 vs FiO2 relation in mechanically ventilated patients without ARDS (n =10) and with mild or moderate ARDS (n =10). In order to explain the dependency of the PaO2/FiO2 on FiO2, shunt fraction and alveolar - arterial oxygen difference ((A-a)DO2) will be determined in these patients.

Objective:

To study the relation between PaO2/FiO2-ratio and FiO2

Study design:

An unblinded, prospective, interventional study

Study population:

Mechanically ventilated patients > 18 years, admitted to the Intensive Care Unit of VU-Medical Center post cardiac surgery without ARDS (n = 10) and with mild to moderate ARDS (n = 10).

Intervention:

Two interventions will be performed:

1. Modulation of FiO2: FiO2 will be reduced to 21% or until peripheral oxygen saturation of 92%, whatever occurs first. Subsequently FiO2 will be increased up to 100%.
2. Withdrawal of blood: Blood will be withdrawn from the indwelling arterial line and pulmonary artery catheter. No catheters will be inserted for the study. The maximum number of time points is 7. At each time point 1.5 ml of blood will be withdrawn from both the arterial and pulmonary artery catheter for blood gas analysis. At the start and the end of the study period 2 additional blood samples of 5 ml each will be drawn. Accordingly, the maximum amount of blood obtained will be less than 50 ml.

Main study parameters/endpoints:

At each level of FiO2 the following parameters will be assessed:

* Arterial blood gas analysis, including SaO2
* Central Venous oxygen saturation and content
* Hemoglobin
* Body temperature
* End tidal CO2
* VO2 and VCO2
* Ventilatory parameters (tidal volume, respiratory rate, Ppeak Paw)
* Hemodynamics (Bloodpressure and Heart Rate)

ELIGIBILITY:
Inclusion Criteria:

All mechanically ventilated patients, admitted to the Intensive Care Unit of VU-Medical Center post cardiac surgery without ARDS and with mild to moderate ARDS. In order to be eligible to participate in this study, a subject must meet all of the following criteria:

* Mechanically ventilated patients
* Stable hemodynamics
* Stable haemoglobin level
* Stable body temperature
* Stable level of sedation
* Pulmonary-Artery and Artery catheter

Exclusion Criteria:

* Incomplete revascularization after CABG
* Cardiac ischemia
* Neurotrauma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-09-01 (Actual); Primary Completion 2020-01-01 (Estimated); Study Completion 2020-08-01 (Estimated)

PRIMARY OUTCOMES:
The effect of FiO2 on the PaO2/FiO2-ratio | 2 hours
  To study the effect of FiO2 on the PaO2/FiO2-ratio in mechanically ventilated patients post cardiac surgery without ARDS and with mild to moderate ARDS

SECONDARY OUTCOMES:
Shunt fraction, arteriovenous oxygen difference and alveolar - arterial oxygen difference | 2 hours
  Shunt fraction, arteriovenous oxygen difference and alveolar - arterial oxygen difference will be determined to explain the relationship between FiO2 and the PaO2/FiO2-ratio

CONTACTS AND LOCATIONS:
Overall Officials: Angelique Spoelstra - de Man, MD, PhD, Principal Investigator — Amsterdam UMC, location VUmc
Locations (1):
- VU University Medical Center, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No